CLINICAL TRIAL: NCT04185844
Title: American Indian Chronic Renal Insufficiency Cohort Study (AI-CRIC Study)
Acronym: AI-CRIC
Status: Recruiting | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 19-159
Record Dates: First submitted 2019-11-22; First posted 2019-12-04 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine serum, plasma, DNA, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite many advances in our understanding of the natural history and progression of chronic kidney disease (CKD) and cardio vascular disease (CVD) in the parent CRIC study over the past 15 years, important questions about key risk factors for these diseases remain unanswered in the AI population. To address this burden of CKD in AI communities Investigators formed a consortium of investigators with extensive experience in conducting research of chronic diseases including diabetes, cardiovascular and kidney disease in AIs of Southwestern US. The proposed CRIC ancillary cohort study of 500 AIs (AI-CRIC) will rapidly improve our understanding of both potential risk factors for CKD progression, as well as the scope of this disease among AIs. This study leverages the current CRIC study and incorporates the planned activities of the next phase of the study - "CRIC 2018" - by implementing contemporary CRIC protocols for kidney and cardiovascular measurement and outcomes.

DETAILED DESCRIPTION:
Investigators will conduct a longitudinal study of a CKD cohort of Southwest AIs to identify unique risk factors for CKD and CVD progression and compare CKD and CVD event rates and risk factors between AI and the populations represented in CRIC. Investigators will establish a specimen bank to support future ancillary studies designed to identify and examine biomarkers associated with the progression of CKD in AIs.

At the Clinic Visit the following will occur:

* weight is measured
* blood pressure and heart rate are recorded
* information about medical history and medication used recently
* blood draw (about ½ cup) for the following tests: CBC (Complete Blood Count), tests of metabolism, and several other heart and kidney tests
* blood pressure in the leg and arm calculated as the Ankle Brachial Index (ABI)
* urine sample collection for kidney function testing
* complete questionnaires about quality of life, diet, mood, thought processes and physical activity.

This visit takes about 1 to 2 hours. Participants will be contacted by telephone six months after the Baseline Visit to ask about recent medical events and medications.

Participants will be asked to return to the center for annual visits during which many but not all of the procedures described above will be conducted.

Additionally, participants will be asked to participate in one of two substudies using remote data collection techniques to identify trajectories of kidney function and cardiovascular risk sub-phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Glomerular Filtration Rate (GFR): eGFR of =>61<80 and microalbuminuria > 30 or eGRF of =<60 (no microalbuminuria required).

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. life expectancy <3 years;
3. institutionalized subjects;
4. End stage renal disease or renal transplant;
5. renal cancer;
6. myeloma;
7. immunosuppression;
8. Polycystic kidney disease;
9. participation in any clinical trial,
10. current pregnancy
11. current incarceration.
12. Appears unlikely or unable to participate in the required study procedures as assessed by the investigator, study coordinator or designee.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Indians at 3 sites.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Slope of the GFR | 5 years
  Primary outcomes regarding Cardio vascular disease will focus on clinical events indicative of ischemic heart disease, CHF, stroke, and peripheral vascular disease supplemented by radiographic evidence of progressive CVD.

SECONDARY OUTCOMES:
Onset of End Stage Renal Disease | 5 years
  The measure is reflected in decline of GFR levels
Significant loss of renal function | 5 years
  The measure is reflected in decline of GFR levels
Composite clinical outcome defined by the occurrence of either 50% decline, or 25 l/min/1.73 m2 decline in GFR from baseline, or onset of ESRD | 5 years
  The composite clinical outcome includes onset of End Stage Renal Disease, Significant loss of renal function or changes in proteinuria over time from baseline
Slope of change in proteinuria over time | 5 years
  The changes in the levels of proteinuria overtime

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Unruh, MD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - NIDDK-Phoenix Epidemiology and Clinical Research, Phoenix, Arizona
  - First Nations Community Health Source, Albuquerque, New Mexico
  - Zuni Health Initiative Center, Black Rock, New Mexico

REFERENCES:
- See also: Chronic Renal Insufficiency cohort study — http://www.cristudy.org/Chronic-Kidney-Disease/Chronic-Renal-Insufficiency-Cohort-Study/about